CLINICAL TRIAL: NCT04891627
Title: Usak University Faculty of Dentistry
Brief Title: Gingival Crevicular IL-34 and CSF-1 Levels in Patients With Periodontitis and Uncontrolled Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: UsakU8
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis; Diabetes
Keywords: Diabetes,; periodontitis; cytokines
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control groups: individuals with clinically healthy gingiva BOP score less than 10% and PD≤3mm
  Interventions: Diagnostic Test: Gingival crevicular fluid
- Periodontitis group: interdental AL ≥5 mm
  Interventions: Diagnostic Test: Gingival crevicular fluid
- Periodontitis with diabetes group: HbA1c ≥6.5%
  Interventions: Diagnostic Test: Gingival crevicular fluid

INTERVENTIONS:
Diagnostic Test: Gingival crevicular fluid — GCF samples were collected in the morning hours 24-48 hours after clinical periodontal measurement.

SUMMARY:
Type 2 diabetes mellitus is a metabolic disorder. There is a bidirectional association between periodontal disease and DM. Currently there is no data relationship between CSF-1 and IL-34, periodontal disease and diabetes.The aim of this study to investigate GCF levels of IL-34 and CSF-1 in periodontitis subjects with diabetes.

DETAILED DESCRIPTION:
Periodontally healthy (H), periodontitis, and periodontitis with diabetes patients, were recruited for this study.

1. Inclusion criteria for H groups: Individuals with clinically healthy gingiva, no attachment and bone loss, and less than 10% bleeding on probing were included.
2. Inclusion criteria for periodontitis groups: Systemically healthy individuals with interdental CAL ≥ 5 mm and PPD ≥ 6 mm were included.
3. Inclusion criteria for periodontitis with diabetes groups: Type 2 diabetes patients with interdental CAL ≥ 5 mm, PPD ≥ 6 mm, and HbA1c ≥ 6.5% were included.

The plaque index (PI), gingival index (GI), presence of bleeding on probing (BOP), PD, and clinical AL were used for clinical periodontal assessments. All assessments were done with a manual probe. GCF samples were obtained and analyzed using an enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* have 20 teeth
* have diabetes .

Exclusion Criteria:

* Individuals have systemic disease
* smokers;
* pregnant
* those using drugs;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals have diabetes and periodontitis
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
It was aimed to compare IL-34 levels by taking gingival crevicular fluid in systemic healthy, periodontitis and diabetic patients with periodontitis groups. | GCF samples taken within the 1. week after the clinical examination of the patient
  GCF was taken interproximal region.

SECONDARY OUTCOMES:
It was aimed to compare CSF-1 levels by taking gingival crevicular fluid in systemic healthy, periodontitis and diabetic patients with periodontitis groups. | GCF samples taken within the 1. week after the clinical examination of the patient
  GCF was taken interproximal region.

CONTACTS AND LOCATIONS:
Overall Officials: ahu dikilitas, Principal Investigator — University of Usak
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

REFERENCES:
- [Derived] Dikilitas A, Karaaslan F, Evirgen S, Ertugrul AS. Gingival crevicular fluid CSF-1 and IL-34 levels in patients with stage III grade C periodontitis and uncontrolled type 2 diabetes mellitus. J Periodontal Implant Sci. 2022 Dec;52(6):455-465. doi: 10.5051/jpis.2106260313. Epub 2022 Apr 12. PMID 36468466